CLINICAL TRIAL: NCT03158675
Title: Fractional Carbon Dioxide Laser Combined With Topical Corticosteroid and Narrow Band Ultraviolet B in Treatment of Stable Vitiligo.
Brief Title: Fractional Carbon Dioxide Laser,Topical Corticosteroid and Narrow Band Ultraviolet B in Treatment of Stable Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MUAAhmed, principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCO2L
Record Dates: First submitted 2017-05-13; First posted 2017-05-18 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Vitiligo
Keywords: fractional co2 laser, topical steroid,UVB narrow band
MeSH Terms: conditions — Vitiligo | interventions — Lasers; Adrenal Cortex Hormones; Steroids; Phototherapy

STUDY DESIGN:
Intervention Model Description: • Methods:-
  -In each patient: The lesions on one side of the body will be randomly allocated to group A, and the lesions on the other side to group B.
  Group A: will be treated with fractional CO2 laser combined with topical corticosteroid and UVB-NB.
  Group B: will be treated with topical corticosteroid and UVB-NB.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fractional co2 laser&topical steroid (Experimental): participant will be compared with one side of the body to the ather side.
  Intervention:
  -Procedure: Fractional carbon dioxide laser.
  -Drug: Topical corticosteroid.
  -Radiation: Ultraviolet B narrow band.
  Interventions: Procedure: fractional carbon dioxide(CO2) laser; Drug: Topical corticosteroid; Radiation: Ultraviolet B narrow band

INTERVENTIONS:
Procedure: fractional carbon dioxide(CO2) laser — -Fractional CO2 laser: Laser sessions will be performed at half month interval and it will be used with a wave length of 10,600nm.
  Other Names: Laser
Drug: Topical corticosteroid — Topical corticosteroid will be applyed twice weekly on both sides for 4 months.
  Other Names: Topical steroid
Radiation: Ultraviolet B narrow band — Ultraviolet B narrow band will be performed (wave length ranged from 300 to 320nm).The sessions will be performed twice weekly for 4 months.
  Other Names: Phototherapy

SUMMARY:
Vitiligo is an acquired disease with a variable course. It is characterized clinically by well-defined depigmented macules or patches thought to occur secondary to melanocyte dysfunction and loss. it is the most common depigmentation disorder, affecting approximately 0.5 to 2.0 percent of the population and has no predilection for gender or race .

DETAILED DESCRIPTION:
Vitiligo is primarily a clinical diagnosis without the need for diagnostic tools. It classified into three types: segmental vitiligo , nonsegmental vitiligo , and unclassifiable vitiligo .

Onset and disease course may vary by subtype .Although the disease is typically asymptomatic and non-fatal; the profound cosmetic disfigurement it produces has a significant negative impact on the patient's quality of life .

Vitiligo occurs due to a complex interaction among genetic, environmental and immunologic factors. This ultimately leads to melanocyte damage resulting characteristic depigmented lesions.

Conventional vitiligo treatments include topical steroid, topical and oral immunomodulators and phototherapy. In spite of much advancement in pharmacotherapy, treatment for vitiligo still remains a challenge for physicians. Re-pigmentation of the lesions on the extremities or over bony prominences is particularly poor due to the reduced numbers of follicle-based melanocytes in these areas .

Treatment of vitiligo with narrowband ultraviolet B light is an important component of the current standard of care.Narrowband ultraviolet B therapy or topical corticosteroid has long been used in vitiligo. However, the re-pigmentation is always transient and time-consuming .

Using surgical therapies (Dermabrasion) may increase the rate of re-pigmentation or erbium-doped yttrium aluminum garnet laser to stimulate melanocyte stem cells and enhance drug absorption and autoinoculation of melanocytes from the margin, but create wounds that take a longer time to heal . In addition to being costly and time consuming, special training, staff, and equipment are needed in order to perform the procedures.

Fractional carbon dioxide lasers, originally developed for tissue rejuvenation and scar remodeling. Recently, it has been used in the treatment of vitiligo. The newly developed fractional carbon dioxide laser does not ablate the entire epidermis, leaving intact skin between coagulated necrotic columns. It decreases risk of potential side effects and minimizes duration of sick leave.

Several mechanisms may contribute to explain the improvement of Vitiligo after fractional carbon dioxide laser sessions. Firstly, wounding therapies may regenerate de novo hair follicles by Wnt-dependant pathway .Moreover the role of hair follicles in the repigmentation of Vitiligo is longstanding knowledge . Secondly, wounding therapies and fractional wounding-therapies may increase the penetration and the well-known efficiency of ultraviolet-radiation. Thirdly, they may induce the activation, proliferation and migration of melanoblasts from the border areas or differentiation of stem cells from the dermis of lesions by initiating propigmenting cytokinic inflammatory cascades .

Adding fractional carbon dioxide laser treatment to the conventional therapies of vitiligo may improve repigmentation rate as well as patient satisfaction .

Aim of the Work :

To evaluate the use of fractional Co2 laser combined with topical corticosteroid and ultraviolet B narrow band( UVB-NB) in treatment of stable vitiligo.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 14 years old.
* Any sex

Exclusion Criteria:

* Patients less than 14 years old.
* Patients with new, spreading lesions of vitiligo within the preceding 6 months.
* Pregnant female patients.
* Patients with history of keloid formation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
VASI scor-Vitiligo Area and Severity Index: | 4 months
  Vitiligo Area and Severity Index (VASI) One hand unit ,which encompasses the palm plus the volar surface of all the digits,is approximately 1% of the total body surface area and is used as a guide to estimate the baseline percentage of vitiligo involvement in each body region.The body is divided into five separate and mutually exclusive regions: hands ,upper extremities (excluding hands),trunk,lower extremities(excluding feet),and feet.The axillary region is included with the upper extremities while the buttocks and inguinal areas are included with the lower extremities.The extent of residual depigmentation is expressed by the following percentages:0,10%,25%,50%,75%,90%,or100%.At 100% depigmentation,no pigment is present; at 90%,specks of pigment is present; at75%,the depigmented area exceeds the pigmented area; at50%,the depigmented and pigmented area are equal; at 25%,the pigmented area exceeds the depigmented area; at10% only specks of depigmentation are present.

SECONDARY OUTCOMES:
Scoring system of repigmentation | 4 months
  * G0,<25% repigmentation (poor)
  * G1,25-50% repigmentation (fair)
  * G2,50-75% repigmentation (good)
  * G3,>75% repigmentation (excellent).
Patient satisfaction | 4 months
  * 0 - not satisfactory
  * to 10 - very satisfactory

CONTACTS AND LOCATIONS:
Overall Officials: Muna Abdullah, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayoumi W, Fontas E, Sillard L, Le Duff F, Ortonne JP, Bahadoran P, Lacour JP, Passeron T. Effect of a preceding laser dermabrasion on the outcome of combined therapy with narrowband ultraviolet B and potent topical steroids for treating nonsegmental vitiligo in resistant localizations. Br J Dermatol. 2012 Jan;166(1):208-11. doi: 10.1111/j.1365-2133.2011.10564.x. Epub 2011 Nov 17. PMID 21824124
- [Background] Beachkofsky TM, Henning JS, Hivnor CM. Induction of de novo hair regeneration in scars after fractionated carbon dioxide laser therapy in three patients. Dermatol Surg. 2011 Sep;37(9):1365-8. doi: 10.1111/j.1524-4725.2011.01934.x. Epub 2011 Apr 14. No abstract available. PMID 21492302
- [Background] Benzekri L, Ezzedine K, Gauthier Y. Vitiligo Potential Repigmentation Index: a simple clinical score that might predict the ability of vitiligo lesions to repigment under therapy. Br J Dermatol. 2013 May;168(5):1143-6. doi: 10.1111/bjd.12147. Epub 2013 Mar 7. No abstract available. PMID 23464539
- [Background] Cui J, Shen LY, Wang GC. Role of hair follicles in the repigmentation of vitiligo. J Invest Dermatol. 1991 Sep;97(3):410-6. doi: 10.1111/1523-1747.ep12480997. PMID 1714927
- [Background] Dillon AB, Sideris A, Hadi A, Elbuluk N. Advances in Vitiligo: An Update on Medical and Surgical Treatments. J Clin Aesthet Dermatol. 2017 Jan;10(1):15-28. Epub 2017 Jan 1. PMID 28210378
- [Background] Ezzedine K, Lim HW, Suzuki T, Katayama I, Hamzavi I, Lan CC, Goh BK, Anbar T, Silva de Castro C, Lee AY, Parsad D, van Geel N, Le Poole IC, Oiso N, Benzekri L, Spritz R, Gauthier Y, Hann SK, Picardo M, Taieb A; Vitiligo Global Issue Consensus Conference Panelists. Revised classification/nomenclature of vitiligo and related issues: the Vitiligo Global Issues Consensus Conference. Pigment Cell Melanoma Res. 2012 May;25(3):E1-13. doi: 10.1111/j.1755-148X.2012.00997.x. PMID 22417114
- [Background] Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI)--a simple practical measure for routine clinical use. Clin Exp Dermatol. 1994 May;19(3):210-6. doi: 10.1111/j.1365-2230.1994.tb01167.x. PMID 8033378
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] Ito M, Yang Z, Andl T, Cui C, Kim N, Millar SE, Cotsarelis G. Wnt-dependent de novo hair follicle regeneration in adult mouse skin after wounding. Nature. 2007 May 17;447(7142):316-20. doi: 10.1038/nature05766. PMID 17507982
- [Background] Li L, Wu Y, Li L, Sun Y, Qiu L, Gao XH, Chen HD. Triple combination treatment with fractional CO2 laser plus topical betamethasone solution and narrowband ultraviolet B for refractory vitiligo: a prospective, randomized half-body, comparative study. Dermatol Ther. 2015 May-Jun;28(3):131-4. doi: 10.1111/dth.12202. Epub 2015 Mar 5. PMID 25753514
- [Background] Mulekar SV, Isedeh P. Surgical interventions for vitiligo: an evidence-based review. Br J Dermatol. 2013 Oct;169 Suppl 3:57-66. doi: 10.1111/bjd.12532. PMID 24098901
- [Background] Salman A, Kurt E, Topcuoglu V, Demircay Z. Social Anxiety and Quality of Life in Vitiligo and Acne Patients with Facial Involvement: A Cross-Sectional Controlled Study. Am J Clin Dermatol. 2016 Jun;17(3):305-11. doi: 10.1007/s40257-016-0172-x. PMID 26818062
- [Background] Vachiramon V, Chaiyabutr C, Rattanaumpawan P, Kanokrungsee S. Effects of a preceding fractional carbon dioxide laser on the outcome of combined local narrowband ultraviolet B and topical steroids in patients with vitiligo in difficult-to-treat areas. Lasers Surg Med. 2016 Feb;48(2):197-202. doi: 10.1002/lsm.22389. Epub 2015 Jul 14. PMID 26175036